CLINICAL TRIAL: NCT01589926
Title: Early Bi-Level Positive Airway Pressure (BiPAP) Ventilation for Acute Chest Syndrome (ACS) - a Double-Blind Randomized Controlled Pilot Study
Brief Title: Bi-Level Positive Airway Ventilation for Acute Chest Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Deepa Manwani, Professor, Pediatrics, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 12-04-139
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Sickle Cell Anemia; Acute Chest Syndrome
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bi-level Positive Airway Pressure Device (Experimental): BiPAP initiated for at least 16 hours per day for a minimum of 48hrs.
  Interventions: Device: Bi-level positive airway pressure device
- Sham CPAP (Sham Comparator): Physiologic continuous positive airway pressure (CPAP) initiated for at least 16 hours per day for a minimum of 48hrs.
  Interventions: Device: Sham CPAP

INTERVENTIONS:
Device: Bi-level positive airway pressure device — BiPAP initiated for at least 16 hours per day for a minimum of 48hrs.
  Arms: Bi-level Positive Airway Pressure Device
Device: Sham CPAP — Sham CPAP initiated for at least 16 hours per day for a minimum of 48hrs.
  Arms: Sham CPAP

SUMMARY:
Acute chest syndrome (ACS) is a frequent complication of sickle cell disease and is diagnosed by having findings on a chest x-ray and one of the following: chest pain, fever, or trouble breathing. Patients with Acute Chest Syndrome can get very sick and require an exchange transfusion (special large blood transfusion) and mechanical ventilation. Bi-level Positive Airway Pressure (also known as BLPAP or BiPAP) is a device that blows air into a patients lungs via a mask that covers the nose. The goal of this study is to determine whether giving children BiPAP when they have ACS, in addition to providing standard clinical care for ACS, alters the clinical course of these patients. The investigators hypothesize that patients receiving effective BiPAP will have milder clinical courses resulting in shorter hospital stays and fewer transfers to the intensive care unit and exchange transfusions.

DETAILED DESCRIPTION:
Acute chest syndrome (ACS) is a frequent complication of sickle cell disease and is diagnosed by a new infiltrate on chest x-ray and one of the following: chest pain, fever, or respiratory signs or symptoms (tachypnea, cough, new onset hypoxemia, or increased work of breathing.)The treatment for acute chest syndrome is focused on supportive care with hydration, antibiotics, blood transfusions and respiratory support. Unfortunately, despite these treatments many patients fail to have improvements in their respiratory status, or have respiratory decompensation. These patients require more aggressive treatments, which frequently include exchange transfusions, pediatric intensive care unit (PCCU) management, and respiratory support.

The study objective is to perform a prospective double blind randomized control trial to investigate if early initiation of effective BiPAP in addition to providing standard clinical care for ACS alters the clinical course of these patients vs. sham BiPAP and standard clinical care. Investigators hypothesize that participants receiving effective BiPAP will have milder clinical courses resulting in shorter hospital stays and fewer transfers to PCCU and exchange transfusions.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with Hemoglobin SS (HB SS), the most common type of sickle cell disease
* patients diagnosed with Hemoglobin SC (HB SC), the second most common type of sickle cell disease.
* patients diagnosed with Hemoglobin sickle beta-zero thalassemia ( HB SB0thal) or Hemoglobin sickle thalassemia (HB SBthal)

Must meet clinical criteria for ACS- an infiltrate on Chest X-ray and one of the following:

* Respiratory symptoms/signs (patients pulse oximetry < 92% or oxygen saturation < 2% below their baseline, tachypnea, cough, and increased work of breathing)
* Fever
* Chest pain AND

Patients' eligible for a simple transfusion based on one of the following criteria:

* Hypoxemia (patients pulse oximetry < 92% or oxygen saturation < 2% below their baseline)
* Hemoglobin < 5 gm/dl
* Increased work of breathing

Exclusion Criteria:

* Patient requires exchange transfusion within first 24 hours of admission
* Patient requires PCCU transfer within first 24 hours of admission
* Hemoglobin > 9gm/dl secondary to these patients requiring an exchange transfusion

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Manwani, MD, Principal Investigator — Albert Einstein College of Medicine; Michael E Roth, MD, Principal Investigator — Albert Einstein College of Medicine; Kerry Morrone, MD, Study Director — Albert Einstein College of Medicine; Hiren Muzumdar, MD, Principal Investigator — Albert Einstein College of Medicine; Ranaan Arens, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Children's Hospital @ Montefiore, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Groups:
- Bi-level Positive Airway Pressure: BiPAP initiated for at least 16 hours per day for a minimum of 48hrs.
  Bi-level positive airway pressure device: BiPAP initiated for at least 16 hours per day for a minimum of 48hrs.
- Sham CPAP: Physiologic CPAP initiated for at least 16 hours per day for a minimum of 48hrs.
  Sham CPAP: Sham CPAP initiated for at least 16 hours per day for a minimum of 48hrs.
Period: Overall Study
Arm/Group | Bi-level Positive Airway Pressure | Sham CPAP
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bi-level Positive Airway Pressure | Sham CPAP | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay as Measured by the Time From Initial Diagnosis of ACS Until Meeting Discharge Criteria.
Description: Length of stay as measured by the time from initial diagnosis of ACS until meeting discharge criteria. It is anticipated length of stay will correlate to efficacy of treatment: shorter stay is theorized to indicate more efficient treatment.
Time Frame: From diagnosis of ACS until meeting discharge criteria- Average 7 days.
Population: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Arm/Group | Bi-level Positive Airway Pressure | Sham CPAP
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Rate of Exchange Transfusions.
Time Frame: Diagnosis until discharge. Average 7 days.
Population: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Arm/Group | Bi-level Positive Airway Pressure | Sham CPAP
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Determine Parent and Patient Acceptability of BLPAP Administration in the Setting of ACS.
Time Frame: Upon completion of intervention at 48hrs.
Population: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Arm/Group | Bi-level Positive Airway Pressure | Sham CPAP
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Rate of PCCU Transfers.
Time Frame: Diagnosis until discharge. Average 7 days.
Population: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Arm/Group | Bi-level Positive Airway Pressure | Sham CPAP
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Difference in Respiratory Rate.
Time Frame: 48hrs after initiation of treatment
Population: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Arm/Group | Bi-level Positive Airway Pressure | Sham CPAP
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Difference in Pulmonary Function Tests.
Time Frame: 48hrs after initiation of treatment
Population: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Arm/Group | Bi-level Positive Airway Pressure | Sham CPAP
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Difference in Mean SpO2 Recording During Sleep.
Description: Peripheral capillary oxygen saturation (SpO2) is an estimate of the amount of oxygen in the blood. It is the percentage of haemoglobin containing oxygen compared to the total amount of haemoglobin in the blood (i.e. oxygenated haemoglobin vs oxygenated and non-oxygenated haemoglobin).
Time Frame: 48hrs after initiation of treatment
Population: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Arm/Group | Bi-level Positive Airway Pressure | Sham CPAP
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Description: Study was terminated due to low enrollment. Only three participants were enrolled and none initiated treatment.
Arm/Group | Bi-level Positive Airway Pressure | Sham CPAP
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes